CLINICAL TRIAL: NCT01847495
Title: Prospective Evaluation of Low-dose Irinotecan and Cyberknife® Stereotactic Body Radiotherapy in the Treatment of Patients With Colorectal Cancer and Limited Liver Metastasis
Brief Title: Evaluation of Low-dose Irinotecan and Cyberknife® SBRT to Treat Colorectal Cancer With Limited Liver Metastasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5443
Record Dates: First submitted 2013-04-12; First posted 2013-05-07 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer
Keywords: Stage IV Colorectal Carcinoma; Liver metastasis; Cyberknife; Stereotactic Body Radiotherapy; SBRT; Irinotecan HCl; CPT-11
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-Dose Irinotecan & CyberKnife SBRT (Experimental): Irinotecan 40mg/m2 x 3-5 days + CyberKnife SBRT 45-60Gy x 3-5 fractions
  Interventions: Drug: Irinotecan; Radiation: CyberKnife

INTERVENTIONS:
Drug: Irinotecan — 40mg/m2 x 3-5 days
  Other Names: Camptosar; Irinotecan Hydrochloride; Irinotecan HCl; CPT-11
Radiation: CyberKnife — 45-60 Gy for 3-5 days CyberKnife SBRT to liver metastasis within 10 elapsed days. Irinotecan will be administered on the same day, prior to SBRT.
  Other Names: Stereotactic Radiosurgery

SUMMARY:
The purpose of this study is to determine the effects of CyberKnife stereotactic body radiotherapy in combination with irinotecan chemotherapy in patients with colon or rectal cancer that has spread to the liver.

Conventional radiation therapy has a limited role in the treatment of patients with liver metastases because the radiation doses are limited by liver toxicity. The CyberKnife system is a type of radiation machine that precisely focuses large doses of x-rays on the tumor, so that injury from radiation to the nearby normal tissue will be minimal. It is approved by the U.S. Food and Drug Administration to treat tumors, lesions and conditions anywhere in the body when radiation therapy is required. While the device is no longer classified as "investigational", the best treatment dose and times are still being evaluated.

Chemotherapy delivered with radiation therapy can increase the effectiveness of treatment, and may allow for a lower dose of radiation therapy to be utilized, thereby limiting negative side effects.

In this study, patients will receive Cyberknife radiosurgery directed to liver metastasis for 3-5 treatments, given every other day. Irinotecan 40mg/m2 will be administered intravenously daily for 3-5 days (5 treatments within 10 elapsed days), and prior to radiation therapy. Patients will have follow-up visits at months 1,2,4,6,9,12,15,18, 24, 30, 36, and every 6 months thereafter for 3 years.

ELIGIBILITY:
* Age>18 years
* Histologically confirmed primary colorectal cancer
* Stage IV colorectal cancer with </= 3 metastases, up to 5cm in size.
* CT scan or MRI of the abdomen with contrast, 60days prior to enrollment
* If patient is allergic to contrast, imaging without contrast is acceptable
* Positron-Emission Tomography 60 days prior to enrollment
* No additional sites of metastasis at the time of protocol enrollment. History of other sites of metastasis that are currently controlled are acceptable.
* No malignant ascites
* At least 4 weeks from any chemotherapy
* No prior liver radiation therapy
* ECOG performance status 0-1
* Life expectancy>3months
* Laboratory evaluations completed 60 days prior to treatment including CMP, CBC with differential, liver function test, and prothrombin time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events related to toxicities from concurrent SBRT and irinotecan | 3 years

SECONDARY OUTCOMES:
Tumor response rate | 3 years
Progression free survival | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Arica Hirsch, MD, Study Chair — Advocate Lutheran General Hospital; James Ruffer, MD, Study Chair — Advocate Lutheran General Hospital; Jacob Bitran, MD, Study Chair — Advocate Lutheran General Hospital; Edward S James, M.D., Study Chair — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States